CLINICAL TRIAL: NCT05496348
Title: Early therapeUtic RespOnse and Predictivity of Long-term Effectiveness of Upadacitinib in Ulcerative Colitis (EUROPE)
Brief Title: Study of Oral Upadacitinib to Assess Change in Disease Activity in Adult Participants With Ulcerative Colitis
Acronym: EUROPE
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-430
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; UC; Upadacitinib; UPA; RINVOQ
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Upadacitinib: Participants will receive upadacitinib as prescribed by their physician according to local label

SUMMARY:
Ulcerative colitis (UC) is a type of inflammatory bowel disease that causes inflammation and bleeding from the lining of the rectum and colon (large intestine).This study will assess how effective upadacitinib is in treating UC.

Upadacitinib (RINVOQ) is an approved drug for treating UC. Approximately 400 adult participants who are prescribed Upadacitinib by their physician in accordance with local label will be enrolled in Germany, Austria and Switzerland.

Upadacitinib will be administered in accordance with the terms of the local marketing authorization, and treatment of participants will be determined solely by the investigator. Participants in the study will be followed for up to 2 years.

There will be no additional burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and only data which are routinely collected during a regular visit will be utilized for this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with an endoscopically confirmed diagnosis of active moderate to severe Ulcerative colitis (UC).
* Participants initiating Upadacitinib (UPA) at the investigator's discretion as part of their routine clinical care; the decision to administer UPA must be made prior to and independent of documentation for the study and according to the approved local label.
* Participants able to understand and communicate with the investigator and comply with the requirements of the study.
* Participants willing to continue with study documentation after cessation of UPA.

Exclusion Criteria:

* Participants with any contraindication to Upadacitinib (UPA).
* Participants previously exposed to a Janus kinase (JAK) inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with Ulcerative colitis (UC)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving symptomatic remission per partial adapted Mayo score among those who achieved clinical response and/or intestinal ultrasound (IUS) response at week 8 of upadacitinib (UPA) induction | Week 52
  Symptomatic remission per partial adapted Mayo score is defined as stool frequency (SF)=0/1 and rectal bleeding score (RBS) =0.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (94):
- Austria (3):
  - Kepler Universitaetsklinikum GmbH /ID# 251868, Linz, Upper Austria
  - Krankenhaus der Barmherzigen Brueder Wien /ID# 251867, Vienna, Vienna
  - Krankenhaus der Barmherzigen Brueder Salzburg /ID# 251869, Salzburg
- Germany (86):
  - Universitaetsklinik Heidelberg /ID# 249922, Heidelberg, Baden-Wurttemberg
  - Praxis fuer Gastroenterologie /ID# 249917, Heidelberg, Baden-Wurttemberg
  - Rems-Murr-Klinikum Winnenden /ID# 278791, Winnenden, Baden-Wurttemberg
  - Klinikum Augsburg /ID# 249979, Augsburg, Bavaria
  - Medizinisches Versorgunszentrum Dachau /ID# 249945, Dachau, Bavaria
  - TUM Klinikum rechts der Isar /ID# 262176, Munich, Bavaria
  - Dr.med. Johannes Behrendt Facharzt für Innere Medizin und Gastroenterologie /ID# 260516, Brandenburg, Brandenburg
  - Praxis Dr. Grümmer /ID# 249925, Potsdam, Brandenburg
  - Private Practice - Dr. Kempelmann /ID# 249935, Tostedt, Hamburg
  - Klinikum Darmstadt /ID# 267685, Darmstadt, Hesse
  - Praxis Dres. Hurst/Simonis /ID# 255421, Darmstadt, Hesse
  - Interdisziplinaeres Crohn Colitis Zentrum /ID# 252622, Frankfurt am Main, Hesse
  - Bethanien-Krankenhaus /ID# 260865, Frankfurt am Main, Hesse
  - Gastroenterologie Opernstrasse Private Practice - Dr. Falk & Krause & Kuhn /ID# 251822, Kassel, Hesse
  - Mueller/Mueller-Ziehm, Hanover /ID# 252617, Hanover, Lower Saxony
  - Medizinische Hochschule Hannover /ID# 254980, Hanover, Lower Saxony
  - Klinikum Lueneburg /ID# 249948, Lüneburg, Lower Saxony
  - Verein für Wissenschaft und Forschung /ID# 249928, Oldenburg, Lower Saxony
  - Private Practice - Dr. Mechthild Kemper & Dr. Markus Dreck /ID# 249916, Coesfeld, North Rhine-Westphalia
  - Evangelisches Krankenhaus Kalk /ID# 249987, Cologne, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis Herne /ID# 249990, Herne, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis Minden /ID# 249914, Minden, North Rhine-Westphalia
  - Dres. Mallach/Spelter /ID# 270912, Wuppertal, North Rhine-Westphalia
  - Benner & Dommermuth /ID# 249896, Koblenz, Rhineland-Palatinate
  - St. Marien- und St. Annastiftskrankenhaus /ID# 273172, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Klinikum Worms gGmbH /ID# 269804, Worms, Rhineland-Palatinate
  - Gemeinschaftspraxis Drs. Denger und Pfitzner /ID# 249974, Friedrichsthal, Saarland
  - Zentrum für Gastroenterologie Saar MVZ GmbH /ID# 249971, Saarbrücken, Saarland
  - Klinikum Chemnitz - Flemmingstraße /ID# 259156, Chemnitz, Saxony
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 249989, Dresden, Saxony
  - Private Practice - Dr. Johannes Janschek /ID# 255092, Dresden, Saxony
  - Universitaetsklinikum Leipzig /ID# 262612, Leipzig, Saxony
  - Gesellschaft für klinische Studien /ID# 254081, Leipzig, Saxony
  - Praxisgemeinschaft Jerichow Schulze /ID# 262931, Jerichow, Saxony-Anhalt
  - Gemeinschaftspraxis im Medicum /ID# 249930, Altenholz, Schleswig-Holstein
  - Praxis S. Tetzlaff /ID# 253770, Buedelsdorf, Schleswig-Holstein
  - Thormann and Bethge /ID# 249897, Kiel, Schleswig-Holstein
  - Gastroenterologisch - Hepatologisches MVZ Kiel GmbH /ID# 252623, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Schleswig-Holstein Campus Luebeck /ID# 249984, Lübeck, Schleswig-Holstein
  - Praxis fuer Gastroenterologie /ID# 249907, Lübeck, Schleswig-Holstein
  - Friedrich-Ebert-Krankenhaus GmbH /ID# 249973, Neumünster, Schleswig-Holstein
  - Gemeinschaftspraxis Dr. med. Maik Weisflog Dr. med. Katrin Ende /ID# 249918, Erfurt, Thuringia
  - Universitaetsklinikum Jena /ID# 253768, Jena, Thuringia
  - Universitaetsklinikum Jena /ID# 254371, Jena, Thuringia
  - Praxis Dr. Schiffelholz /ID# 252621, Augsburg
  - MVZ Gastro Friedrichshain /ID# 249924, Berlin
  - Praxis Dr. Berndt /ID# 252067, Berlin
  - Dres. Schick/Wesenberg /ID# 249977, Berlin
  - MVZ fuer Gastroenterlogie am Bayerischen Platz /ID# 249981, Berlin
  - Zweite Gemeinnuutzige Krankenhaus GmbH DRK Kliniken Berlin Kopenick /ID# 262849, Berlin
  - Praxis S. Grüngreiff /ID# 249927, Berlin
  - Praxis Dr. Soellenboehmer /ID# 249985, Berlin
  - Praxis Dr. Spitz /ID# 252616, Berlin
  - Krankenhaus Waldfriede /ID# 249900, Berlin-Zehlendorf
  - Internist. Facharztp. Dr. Palmai /ID# 251821, Bitterfeld-Wolfen
  - Alb-Donau Klinikum Blaubeuren, ADK GmbH für Gesundheit und Soziales /ID# 249923, Blaubeuren Abbey
  - Frach/Hohaus, Dresden, DE /ID# 254979, Dresden
  - Dres. Krause/Schiffer /ID# 251727, Frechen
  - Dres. Bauer/Doerflinger /ID# 251568, Freiburg im Breisgau
  - Internisten in Geldern /ID# 252068, Guelders
  - Universitaetsklinikum Halle (Saale) /ID# 254083, Halle
  - Private Practice - Dr. Matthias Eichler /ID# 249933, Hamburg
  - Tappe/Miks/Delker, Hamm, DE /ID# 251729, Hamm
  - Internistische Praxisgemeinschaft Hanau GbR /ID# 254079, Hanau
  - Gastroenterologische Gemeinschaftspraxis /ID# 263633, Heilbronn
  - Städtisches Kh. Heinsberg GmbH /ID# 252624, Heinsberg
  - Praxis Dres. Preiss/Engelke /ID# 249919, Herne
  - Praxis Dr. Schwarz /ID# 251819, Hettstedt
  - MVZ Dres. Al-Kadi & Partner /ID# 249929, Iserlohn
  - Praxis Dr. Weber /ID# 256099, Jena
  - Gastroenterologe am Ettlinger Tor /ID# 249982, Karlsruhe
  - MVZ Doceins West GmbH /ID# 249915, Koblenz
  - MVZ Gastroenterologie Leverkusen /ID# 260512, Leverkusen
  - Gastropraxis Magdeburg /ID# 249988, Magdeburg
  - Praxis Dr. Burlefinger /ID# 259159, Munich
  - Prof-med-stud.de /ID# 255419, Munich
  - Medizinisches Versorgungszentrum Portal 10 /ID# 249947, Münster
  - Gastro Campus Research GbR /ID# 249983, Münster
  - Praxis Dres Brendel /ID# 254078, Nuremberg
  - Medius Klinik Nürtingen /ID# 255420, Nürtingen
  - Pc Docs /Id# 249921, Pirmasens
  - Elisabeth Klinikum GmbH /ID# 252264, Schmalkalden
  - Praxis fuer Gastroenterologie /ID# 252615, Schwerin
  - Dres. Rehbehn/Skusa /ID# 252618, Solingen
  - bauchraum Gastroenterologisches Zentrum Dres. F. Kuehl, C. Hartmann, T. Klag BAG /ID# 251567, Stuttgart
  - Dr. Schirin-Sokhan /ID# 259158, Würselen
- Switzerland (5):
  - Zentrum fur Gastroenterologie und Hepatologie /ID# 260967, Zurich, Canton of Zurich
  - University Hospital Zurich /ID# 260966, Zurich, Canton of Zurich
  - EOC Ospedale Regionale Lugano /ID# 277165, Lugano, Canton Ticino
  - Inselspital, Universitaetsspital Bern /ID# 260968, Bern
  - Berner IBD Study Group /ID# 262315, Bern

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related info — https://www.rxabbvie.com/